CLINICAL TRIAL: NCT01748799
Title: Effects of Fixed or Self-Titrated Dosages of Sativex on Cannabis Users
Brief Title: Fixed or Self-Titrated Dosages of Sativex on Cannabis Users
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre for Addiction and Mental Health (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government)
Responsible Party: Principal Investigator, Bernard Le Foll, Head, Translational Addiction Research Laboratory, Centre for Addiction and Mental Health
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: 103/2011; 243152 (Other Grant/Funding Number: Canadian Institutes of Health Research)
Record Dates: First submitted 2012-12-08; First posted 2012-12-13 (Estimated); Results first posted 2016-02-01 (Estimated); Last update posted 2016-02-01 (Estimated); Status verified 2015-10

CONDITIONS: Cannabis Dependence
Keywords: Cannabis dependence; Sativex
MeSH Terms: conditions — Marijuana Abuse | interventions — nabiximols; Dronabinol; Cannabidiol; Ethanol; Propylene Glycol; peppermint oil; Color

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (8):
- Sequence 1 (Other): Self-titrated placebo - Self-titrated Sativex - Fixed dose Sativex - Fixed dose placebo
  Interventions: Drug: Sativex; Drug: Placebo
- Sequence 2 (Other): Fixed dose placebo - Fixed dose Sativex - Self-titrated Sativex - Self-titrated placebo
  Interventions: Drug: Sativex; Drug: Placebo
- Sequence 3 (Other): Fixed dose placebo - Fixed dose Sativex - Self-titrated placebo - Self-titrated Sativex
  Interventions: Drug: Sativex; Drug: Placebo
- Sequence 4 (Other): Fixed dose Sativex - Fixed dose placebo - Self-titrated placebo - Self-titrated Sativex
  Interventions: Drug: Sativex; Drug: Placebo
- Sequence 5 (Other): Self-titrated Sativex - Self-titrated placebo - Fixed dose Sativex - Fixed dose placebo
  Interventions: Drug: Sativex; Drug: Placebo
- Sequence 6 (Other): Self-titrated Sativex - Self-titrated placebo - Fixed dose placebo - Fixed dose Sativex
  Interventions: Drug: Sativex; Drug: Placebo
- Sequence 7 (Other): Self-titrated placebo - Self-titrated Sativex - Fixed dose placebo - Fixed dose Sativex
  Interventions: Drug: Sativex; Drug: Placebo
- Sequence 8 (Other): Fixed dose Sativex - Fixed dose placebo - Self-titrated Sativex - Self-titrated placebo
  Interventions: Drug: Sativex; Drug: Placebo

INTERVENTIONS:
Drug: Sativex — All participants received the same interventions (Fixed or Self-Titrated Sativex), just in different sequences.
  Other Names: Delta-9-tetrahydrocannabinol and cannabidiol
Drug: Placebo — All participants received the same interventions (Fixed or Self-Titrated Placebo), just in different sequences.
  Other Names: Ethanol, propylene glycol and peppermint oil with colors

SUMMARY:
The purpose of this study is to to demonstrate the feasibility and tolerability of the use of Sativex in cannabis dependent individuals and to assess the effects of fixed or self titrated dosages of SATIVEX® (Δ9-tetrahydrocannabinol /cannabidiol combination in a buccal spray) on withdrawal symptoms, craving scores and cannabis consumption during the study period.

DETAILED DESCRIPTION:
This will be a one year pilot/feasibility study, assessing the effects of fixed or self-titrated dosages of SATIVEX® (Δ9-tetrahydrocannabinol /cannabidiol combination in a buccal spray) on withdrawal from cannabis and craving among cannabis dependent subjects. Subjects in this study will undergo an 8-week double-blind, placebo-controlled trial. Subjects will be regular cannabis-users who are not currently seeking treatment for cannabis dependence. Subjects will participate in each of 8 conditions, lasting 5 weekdays each (an ABACADAE study design); four smoke as usual conditions (SAU) and four cannabis abstinence conditions. During each abstinence condition (B, C, D, E conditions), subjects will be allocated to one condition including self-titration of placebo, fixed dose of placebo, self-titration of SATIVEX (up to a max of 40 sprays per day, equal to 108mg THC) or fixed dose of SATIVEX (40 sprays per day). Each medication phase will be followed by a washout period where individuals will be requested to smoke cannabis as usual (A condition). The experimental conditions will be: type of SATIVEX® spray used (active vs placebo), and titration regimen (fixed or self-titrated). This pilot study will allow us to demonstrate the feasibility of our approach and to determine the sample size to use secondarily for a larger study. Our ultimate goal is to determine optimal conditions to use for a subsequent randomized controlled trial assessing the efficacy of SATIVEX® in treatment of Cannabis dependence among treatment-seeking subjects.

ELIGIBILITY:
Inclusion Criteria:

* age 18-50
* current cannabis dependence
* cannabis as primary drug of abuse
* frequent cannabis use (i.e., at least 5 days per week)
* have experienced at least 2 withdrawal symptoms during previous cessation periods
* cannabis use not for medical purposes (i.e., not a government-licensed medical cannabis user)
* not seeking treatment for cannabis dependence
* willingness to participate in study protocol

Exclusion Criteria:

* meet criteria for any psychiatric disorder requiring psychiatric intervention
* have a history of seizures; c)have known sensitivity to Dronabinol, Cannabidiol, Propylene glycole, Ethanol or peppermint oil (used in Sativex buccal spray
* suffer from an unstable medical condition
* currently have physical dependence on any other drugs (excluding nicotine) that would require medical detoxification
* currently taking psychotropic medication with benefit for any other illness than treatment of insomnia
* pregnant or breast-feeding
* hold a job that involves operating heavy machinery
* currently seeking treatment for cannabis-related problems
* family history of psychotic symptoms

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 16 (Actual)
Dates: Start 2013-02; Primary Completion 2014-09 (Actual); Study Completion 2014-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bernard Le Foll, Principal Investigator — Centre for Addiction and Mental Health
Locations (1):
- Centre for Addiction and Mental Health, Toronto, Ontario, Canada

REFERENCES:
- See also: Information about research at the Centre for Addiction and Mental Health, Canada's largest mental health and addiction teaching hospital, fully affiliated with the University of Toronto, and a PAHO/WHO Collaborating Centre — http://www.camh.net/research

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Sequence 1 | Sequence 2 | Sequence 3 | Sequence 4 | Sequence 5 | Sequence 6 | Sequence 7 | Sequence 8
Started | 6 | 1 | 1 | 2 | 1 | 2 | 2 | 1
Completed SAU of Fixed Dose Placebo | 2 | 1 | 1 | 2 | 1 | 1 | 1 | 1
Completed Fixed Dose Placebo | 2 | 1 | 1 | 2 | 1 | 1 | 1 | 1
Completed SAU of Fixed Dose Sativex | 1 | 1 | 1 | 2 | 1 | 1 | 1 | 1
Completed Fixed Dose Sativex | 1 | 1 | 1 | 2 | 1 | 1 | 1 | 1
Completed SAU of Self-titrated Placebo | 5 | 1 | 1 | 2 | 1 | 2 | 1 | 1
Completed Self-titrated Placebo | 4 | 1 | 1 | 2 | 1 | 2 | 1 | 1
Completed SAU of Self-titrated Sativex | 2 | 1 | 1 | 2 | 1 | 2 | 1 | 1
Completed Self-titrated Sativex | 1 | 1 | 1 | 2 | 1 | 1 | 1 | 1
Completed | 1 | 1 | 1 | 2 | 1 | 1 | 1 | 1
Not Completed | 5 | 0 | 0 | 0 | 0 | 1 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Sequence 1 | Sequence 2 | Sequence 3 | Sequence 4 | Sequence 5 | Sequence 6 | Sequence 7 | Sequence 8 | Total
Number analyzed (Participants) | 6 | 1 | 1 | 2 | 1 | 2 | 2 | 1 | 16
Age, Continuous [Mean (Standard Deviation); unit: years] | 35.7 (8.6) | 24.0 (0.0) | 19.0 (0.0) | 46.5 (6.4) | 36.0 (0.0) | 41.5 (6.4) | 43.0 (5.6) | 22.0 (0.0) | 34.8 (10.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 4
  Male | 4 | 0 | 1 | 2 | 1 | 2 | 1 | 1 | 12
Region of Enrollment [Number; unit: participants]
  Canada | 6 | 1 | 1 | 2 | 1 | 2 | 2 | 1 | 16

OUTCOME MEASURES:

1. Primary Outcome: Feasibility
Description: Feasibility will be assessed by analysing how many participants can be recruited/complete the whole (randomly assigned) experimental sequence with a period of one year.
Time Frame: 12 months
Population: 16 participants were enrolled in the study, 9 participants completed the whole (randomly assigned) experimental sequence
Measure: Number; unit: participants
Arm/Group | Sequence 1 | Sequence 2 | Sequence 3 | Sequence 4 | Sequence 5 | Sequence 6 | Sequence 7 | Sequence 8
Number analyzed (Participants) | 6 | 1 | 1 | 2 | 1 | 2 | 2 | 1
participants | 1 | 1 | 1 | 2 | 1 | 1 | 1 | 1

2. Secondary Outcome: Tolerability of Sativex in Persons That Are Cannabis Dependent
Description: To assess what number of participants might withdrew due non-tolerability of Sativex
Time Frame: 8 weeks
Population: Data from 16 participants enrolled in the study was analyzed, none of the participants withdrew due non-tolerability of Sativex
Measure: Number; unit: participants
Arm/Group | Sequence 1 | Sequence 2 | Sequence 3 | Sequence 4 | Sequence 5 | Sequence 6 | Sequence 7 | Sequence 8
Number analyzed (Participants) | 6 | 1 | 1 | 2 | 1 | 2 | 2 | 1
participants | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

3. Secondary Outcome: Cannabis Withdrawal
Description: Withdrawal symptoms were assessed using the Cannabis Withdrawal Scale (CWS) (Minimum-Maximum Scores 0-190, high scores represent more withdrawal) and Cannabis Withdrawal Checklist (CWC) (Minimum-Maximum Scores 0-48, high scores represent more withdrawal) by establishing comparisons between Sativex/Placebo and Smoke as usual conditions (4 interventions: Fixed Sativex, Fixed Placebo, Self-titrated Sativex, Self-titrated Placebo and 4 corresponding Smoke as usual conditions).
Time Frame: 8 weeks
Population: Only 9 of the 16 participants recruited completed the whole experimental sequence (participants were assigned to 1 of 8 different experimental sequences in a randomized order).
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Fixed Dose Sativex: Participants were requested to abstain from using cannabis and take a fixed dose of Sativex during this condition (40 sprays per day). Each abstinence condition was followed by a smoke as usual condition (SAU).
- Smoke as Usual FS: Smoke as usual condition corresponding to Fixed Sativex
- Self-titrated Sativex: Participants were requested to abstain from using cannabis and self-titrate dosages of Sativex (up to 40 sprays per day) during this condition. Each abstinence condition was followed by a smoke as usual condition (SAU).
- Smoke as Usual StS: Smoke as usual condition corresponding to Self-titrated Sativex
- Fixed Dose Placebo: Participants were requested to abstain from using cannabis and administer a fixed dose of placebo daily (40 sprays per day). Each abstinence condition was followed by a smoke as usual condition (SAU).
- Smoke as Usual FP: Smoke as usual condition corresponding to Fixed Placebo
- Self-titrated Placebo: Participants were requested to abstain from using cannabis and self-titrate dosages of placebo (up to 40 sprays per day) during this condition. Each abstinence condition was followed by a smoke as usual condition (SAU).
- Smoke as Usual StP: Smoke as usual condition corresponding to Self-titrated Placebo
Arm/Group | Fixed Dose Sativex | Smoke as Usual FS | Self-titrated Sativex | Smoke as Usual StS | Fixed Dose Placebo | Smoke as Usual FP | Self-titrated Placebo | Smoke as Usual StP
Number analyzed (Participants) | 9 | 9 | 9 | 9 | 9 | 9 | 9 | 9
units on a scale
  Cannabis Withdrawal Scale (CWS) | 10.3 (12.2) | 7.9 (10.0) | 9.8 (10.9) | 6.6 (5.8) | 17.9 (15.9) | 8.6 (11.4) | 13.7 (14.5) | 7.5 (8.3)
  Cannabis Withdrawal Checklist (CWC) Total | 3.6 (3.5) | 2.6 (2.0) | 4.0 (4.2) | 2.3 (2.2) | 7.4 (5.9) | 3.7 (3.4) | 5.9 (5.5) | 3.0 (1.6)
Statistical Analysis 1: Comparison: Fixed Dose Sativex vs Smoke as Usual FS vs Self-titrated Sativex vs Smoke as Usual StS vs Fixed Dose Placebo vs Smoke as Usual FP vs Self-titrated Placebo vs Smoke as Usual StP; Omnibus analysis for Cannabis Withdrawal Scale (CWS) data was a Repeated measures ANOVA (including all the experimental conditions) followed by pair-wise comparisons. The level for statistical significance was p< 0.05; Test type: Superiority or Other; p < 0.01, ANOVA — The level for statistical significance was p< 0.05
Statistical Analysis 2: Comparison: Fixed Dose Sativex vs Smoke as Usual FS vs Self-titrated Sativex vs Smoke as Usual StS vs Fixed Dose Placebo vs Smoke as Usual FP vs Self-titrated Placebo vs Smoke as Usual StP; Omnibus analysis for Cannabis Withdrawal Checklist (CWC) data was a Repeated measures ANOVA (including all the experimental conditions) followed by pair-wise comparisons. The level for statistical significance was p< 0.05; Test type: Superiority or Other; p = 0.01, ANOVA — The level for statistical significance was p< 0.05

ADVERSE EVENTS:
Time Frame: 8 weeks
Description: Some adverse events were not study-related (e.g. mild cold, tension headache or hot flashes) and some expected side effects, such as nausea, sleep problems or diarrhea, were noted.
Groups:
- Fixed Dose Placebo: Participants were requested to abstain from using cannabis and take a fixed dose of placebo during this condition (40 sprays per day). Each abstinence condition was followed by a smoke as usual condition (SAU).
Arm/Group | Fixed Dose Sativex | Smoke as Usual FS | Self-titrated Sativex | Smoke as Usual StS | Fixed Dose Placebo | Smoke as Usual FP | Self-titrated Placebo | Smoke as Usual StP
Serious Adverse Events (participants affected / at risk) | 0/9 | 0/9 | 0/9 | 0/11 | 0/10 | 0/10 | 0/13 | 0/14
Other Adverse Events (participants affected / at risk) | 5/9 | 1/9 | 7/9 | 3/11 | 5/10 | 5/10 | 9/13 | 9/14
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Fixed Dose Sativex (N=9) | Smoke as Usual FS (N=9) | Self-titrated Sativex (N=9) | Smoke as Usual StS (N=11) | Fixed Dose Placebo (N=10) | Smoke as Usual FP (N=10) | Self-titrated Placebo (N=13) | Smoke as Usual StP (N=14)
Nausea (Gastrointestinal disorders) | 0 (0) | 0 | 3 (3) | 0 | 1 (1) | 0 | 0 (0) | 0
Insomnia (Psychiatric disorders) | 1 (1) | 0 | 1 (1) | 0 | 3 (3) | 0 | 1 (1) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 0 (0) | 0 | 2 (2) | 0 | 0 (0) | 0 | 0 (0) | 4 (4)
Cold (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 | 0 (0) | 0 | 1 (1) | 3 (3) | 3 (3) | 0
Nightmares (Psychiatric disorders) | 0 (0) | 0 | 0 (0) | 1 (1) | 1 (1) | 0 | 0 (0) | 0
Pain in the knee (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 | 1 (1) | 0 | 0 (0) | 0 | 1 (1) | 0 — from an old injury
Scapula pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 | 0 (0) | 0 | 1 (1) | 0 | 0 (0) | 0
Sore foot (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 | 1 (1) | 1 (1) | 0 (0) | 0 | 0 (0) | 0
Sore Throat (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 | 0 (0) | 0 | 0 (0) | 0 | 1 (1) | 0
Headache (General disorders) | 1 (1) | 0 | 0 (0) | 0 | 1 (1) | 1 (1) | 3 (3) | 1 (1)
hot flashes (Blood and lymphatic system disorders) | 1 (1) | 0 | 0 (0) | 0 | 1 (1) | 0 | 1 (2) | 0
Impaired taste sensation of food (General disorders) | 0 (0) | 0 | 0 (0) | 0 | 1 (1) | 0 | 1 (1) | 0
Vertigo (General disorders) | 1 (1) | 0 | 1 (1) | 1 (1) | 1 (1) | 0 | 0 (0) | 0
heartburn (Gastrointestinal disorders) | 0 (0) | 0 | 0 (0) | 0 | 0 (0) | 0 | 2 (2) | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 2 (2) | 0 | 0
Rash (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 2 (2) | 1 (1)
Ringing ears (Ear and labyrinth disorders) | 0 | 1 (1) | 0 | 1 (2) | 0 | 0 | 0 | 0
Low motivation (Psychiatric disorders) | 0 | 0 | 0 | 1 (1) | 0 | 0 | 0 | 0
Dry eyes (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 (1) | 0
Runny nose (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 (1) | 0 | 0 | 0 | 0 (0) | 1 (1)
Ankle pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 (1)
Anxiety (Psychiatric disorders) | 0 | 0 | 0 | 1 (1) | 0 | 0 | 0 | 1 (1)
Feeling drowsy (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 (1) | 1 (1)
Stomach Pain (Gastrointestinal disorders) | 0 | 0 | 0 | 1 (1) | 0 | 0 | 0 | 0

LIMITATIONS AND CAVEATS:
The main limitation is the small sample size. Also our study did not include experimental conditions containing THC alone and CBD alone for comparison. The short duration of the experimental condition is also a limitation.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No